CLINICAL TRIAL: NCT07310784
Title: A Multicenter, Randomized, Controlled, Open-label, Phase II Trial on Autologous Tumor Infiltrating Lymphocyte Injection (LM103 TILs) for the Treatment of Advanced Melanoma
Brief Title: A Phase II Trial of LM103 in Advanced Melanoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou BlueHorse Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LM103-MM-CT02
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Advanced Melanoma
MeSH Terms: interventions — Dacarbazine; Temozolomide; Paclitaxel; Carboplatin; Cisplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LM103 TILs Group (Experimental)
  Interventions: Biological: LM103 TILs Injection
- Chemotherapy Group (Active Comparator): Chemotherapy regimen selected by investigators
  Interventions: Drug: Dacarbazine, temozolomide, paclitaxel, carboplatin/cisplatin

INTERVENTIONS:
Biological: LM103 TILs Injection — Extract, culture and expand tumor-infiltrating lymphocytes from resected tumor tissues in vitro for the manufactur of LM103 TILs injection. After NMA-LD, the subjects received LM103 infusion and followed by IL-2 supportive treatment.
  Arms: LM103 TILs Group
Drug: Dacarbazine, temozolomide, paclitaxel, carboplatin/cisplatin — The subjects will start treatment with a chemotherapy regimen selected by the investigators, including dacarbazine, temozolomide, paclitaxel, carboplatin/cisplatin.
  Arms: Chemotherapy Group

SUMMARY:
A total of 92 subjects with advanced melanoma who met the inclusion criteria will be randomly assigned in a 1:1 ratio to the experimental group and the control group in this phase II trial. The study will be followed up until 24 months after treatment.

ELIGIBILITY:
Inclusion Criteria:

* At the date of signing Informed Consent Form (ICF), 18 ~75 years old, male or female;
* Expected survival time >3 months;
* ECOG performance status 0-1;
* Patients with unresectable recurrent/metastatic melanoma (excluding uveal melanoma) who have failed at least two lines of standard treatment: • Patients need to have failed or be intolerant to PD-1 antibody treatment; • If the BRAF V600 mutation is positive, treatment with BRAF±MEK inhibitors must fail; • If the NRAS mutation is positive, treatment with Tunlametinib must fail;
* Patients have lesions that can be used for surgical resection or biopsy puncture;
* Even after tumor tissue resection/biopsy puncture, there should still be at least one measurable lesion (according to RECIST1.1);
* Patients have sufficient hematology and organ functions;
* Voluntarily sign a written informed consent form (ICF).

Exclusion Criteria:

* A history of other malignant tumors within the past 5 years, excluding malignant tumors that can be expected to heal after treatment (including but not limited to well-treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or ductal carcinoma in situ of the breast treated by radical surgery);
* Adverse reactions caused by previous treatments have not been recovered to grade ≤1(CTCAE V5.0) (excluding alopecia and neurotoxicity, and hypothyroidism, adrenal insufficiency and hypopituitarism that cannot be restored to grade 2 as determined by the investigators for a long time);
* Any immune-related adverse reaction (irAE) with a severity level greater than grade 3 that has occurred during any previous immunotherapy and has been permanently discontinued;
* Have received vaccination within two months prior to signing the ICF, or plan to receive vaccination during the study;
* Have received TIL cell therapy, allogeneic T cell therapy or NK cell therapy within 6 months prior to signing the ICF;
* Have received allogeneic hematopoietic stem cell transplantation or solid organ transplantation in the past;
* Suffering from central nervous system metastases and/or cancerous meningitis. Patients who have received brain metastasis treatment and whose conditions have been stable for at least 6 months, and whose disease progression has been confirmed by imaging examinations within 4 weeks before LM103 reinfusion, may consider participating in this study;
* Suffering from or suspected of having an active autoimmune disease;
* Suffering from a large amount of pleural effusion or ascites with clinical symptoms or requiring symptomatic treatment;
* Patients with current or previous irreversible interstitial lung disease;
* Suffering from serious cardiovascular and cerebrovascular diseases;
* Suffering from an active infection that requires systemic treatment;
* Suffering from infectious diseases such as hepatitis B, hepatitis C, syphilis, AIDS;
* Patients with esophageal or gastric varices requiring immediate intervention (such as ligation or sclerotherapy), or those with a higher risk of bleeding as recommended by the investigator or gastroenterologist or hepatologist, evidence of portal hypertension (including splenomegaly found in imaging examinations), or a history of variceal bleeding must undergo endoscopic assessment within 3 months before enrollment;
* Uncontrolled metabolic disorders, such as diabetes, or other non-malignant organ or systemic diseases or secondary reactions to cancer, can lead to higher medical risks and/or uncertainties in survival assessment;
* Those who are known to be allergic to any component of the investigational drug and the LM103 product formula;
* Women who are pregnant or breastfeeding;
* As determined by the investigators, there are other severe, acute or chronic medical diseases, mental disorders or laboratory abnormalities that may increase the risks related to participation in the study or may interfere with the interpretation of the study results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Estimated)
Dates: Start 2025-12-16 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | Every 6 weeks in the first 6 months after treatment and every 12 weeks from 6 months to 24 months
  PFS confirmed by the Independent Review Committee (IRC) according to RECIST 1.1

SECONDARY OUTCOMES:
Overall survival (OS) | Maximum 24 months
  OS and OS rates in 6, 12, 18, 24 months
PFS | Every 6 weeks in the first 6 months after treatment and every 12 weeks from 6 months to 24 months
  PFS confirmed by the investigators according to RECIST 1.1
Objective Response Rate (ORR) | Every 6 weeks in the first 6 months after treatment and every 12 weeks from 6 months to 24 months
  ORR assessed by IRC and investigators according to RECIST 1.1
Disease Control Rates (DCR) | Every 6 weeks in the first 6 months after treatment and every 12 weeks from 6 months to 24 months
  DCR assessed by IRC and investigators according to RECIST 1.1
Duration of Response (DoR) | Every 6 weeks in the first 6 months after treatment and every 12 weeks from 6 months to 24 months
  DoR assessed by IRC and investigators according to RECIST 1.1
Adverse Events (AEs) | Maximum 24 months
  AEs will be recorded and assessed according to CTCAE Version 5.0

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China